CLINICAL TRIAL: NCT07267650
Title: Analgesic Efficacy of iPACK Block Versus Periarticular Infiltration as an Adjunct to Femoral Triangle Block in Total Knee Arthroplasty: A Prospective, Randomized, Double-Blind, Controlled Trial
Brief Title: iPACK Block vs. Periarticular Infiltration for TKA Pain Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turgutlu State Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANES-TKA-2025-001
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Osteoarthritis, Knee / Osteoarthritis, Hip
Keywords: Total Knee Arthroplasty; TKA; Postoperative Pain; Pain Management; Analgesia; Nerve Block; Femoral Triangle Block; FTB; iPACK block; Local Infiltration Analgesia; Randomized Controlled Trial; Timed Up and Go Test; Straight Leg Raise; Periarticular Infiltration; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis; Agnosia | interventions — Surgeons; Anesthesiologists; Bupivacaine; Epinephrine; Methylprednisolone; Cefazolin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FTB + iPACK Group (n=50) (Active Comparator)
  Interventions: Procedure: FTB; Procedure: IPACK block; Procedure: Sham Intervention 1 (Surgeon); Drug: Bupivacaine %0.25 (isobaric); Drug: Normal Saline (0.9% NaCl)
- FTB + PAI Group (n=50) (Experimental)
  Interventions: Procedure: FTB; Procedure: Sham Intervention 2 (Anesthesiologist); Procedure: PAI (Surgeon); Drug: Bupivacaine %0.25 (isobaric); Drug: Bupivacaine + Adrenaline + Methylprednisolone + Cefazoline; Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Procedure: FTB — All patients will receive an ultrasound-guided Femoral Triangle Block (FTB) with 20 mL of 0.25% Bupivacaine, supplemented by an Anterior Femoral Cutaneous Nerve block with 5 mL of the same solution.
Procedure: IPACK block — Patients will receive an ultrasound-guided real iPACK block with 20 mL of 0.25% Bupivacaine
  Arms: FTB + iPACK Group (n=50)
Procedure: Sham Intervention 1 (Surgeon) — Patients will receive a sham Periarticular Infiltration (PAI) with an equivalent volume of normal saline intraoperatively.
  Arms: FTB + iPACK Group (n=50)
Procedure: Sham Intervention 2 (Anesthesiologist) — Patients will receive a sham iPACK block with an equivalent volume of normal saline preoperatively.
  Arms: FTB + PAI Group (n=50)
Procedure: PAI (Surgeon) — The surgeon intraoperatively administers the standardized PAI cocktail (total volume approx. 50 mL): 24 mL 0.5% Bupivacaine, 0.3 mL Adrenaline (1:1000), 40 mg Methylprednisolone, 1 gr Cefazoline, and 22 mL 0.9% Sodium Chloride. The surgeon will administer the infiltration into the medial, lateral, and posterior quadrants of the knee capsule, specifically sparing the anterior quadrant.
  Arms: FTB + PAI Group (n=50)
Drug: Bupivacaine %0.25 (isobaric) — Used for FTB and iPACK blocks.
Drug: Bupivacaine + Adrenaline + Methylprednisolone + Cefazoline — Used for PAI
  Arms: FTB + PAI Group (n=50)
Drug: Normal Saline (0.9% NaCl) — Used for sham/placebo infiltration or block.

SUMMARY:
This study aims to compare two different multimodal analgesic techniques for pain management after total knee arthroplasty (TKA). The primary purpose is to determine if a combination of two specific nerve blocks administered by an anesthesiologist (Femoral Triangle Block + iPACK block) results in superior pain control compared to a combination of a nerve block and a local infiltration administered by the surgeon (FTB + Periarticular Infiltration [PAI]).

The hypothesis is that the FTB + iPACK combination will lead to a significant reduction in Numeric Rating Scale (NRS) pain scores with movement at 24 hours postoperatively.

This will be a prospective, randomized, double-blind, parallel-group, single-center study involving patients scheduled for primary unilateral TKA. Participants will be randomly assigned to one of two groups. All patients, clinicians (anesthesiologists and surgeon), and outcome assessors will be blinded to the group allocation using a double-dummy technique.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a highly successful procedure for end-stage knee osteoarthritis but is associated with significant postoperative pain. Effective pain management is crucial for facilitating early rehabilitation and improving patient comfort. Modern pain management relies on multimodal, opioid-sparing protocols that often include motor-sparing regional anesthesia techniques like the femoral triangle block (FTB).

While FTB provides excellent analgesia for the anterior part of the knee, pain originating from the posterior knee capsule remains a significant challenge. This posterior pain is commonly managed either by the surgeon through a diffuse periarticular infiltration (PAI) of a local anesthetic cocktail or by the anesthesiologist through a targeted, ultrasound-guided block of the posterior capsule known as the iPACK block.

It is currently unclear whether a fully anesthesiologist-driven, neuroanatomically targeted approach (FTB + iPACK) offers superior outcomes compared to a hybrid approach involving both the anesthesiologist and the surgeon (FTB + PAI).

This prospective, randomized, double-blind controlled trial is designed to compare these two advanced analgesic combinations. All patients will receive a standardized spinal anesthetic (3 mL of 0.5% heavy bupivacaine). The study will evaluate which method provides better pain control, measured primarily by Numeric Rating Scale (NRS) pain scores at 24 hours, and secondarily by total rescue analgesic (tramadol) consumption, functional recovery (Timed Up and Go test and Straight Leg Raise test), and knee range of motion.

Sample size will be determined based on an internal pilot study. An initial 30 patients (15 per group) will be enrolled. The mean and standard deviation of the primary outcome (NRS pain score with movement at 24 hours) from this pilot cohort will be used to calculate the final sample size required to detect a clinically significant difference (e.g., 1 point on the NRS) with 80% power and an alpha of 0.05. The final enrollment target is estimated to be approximately 100 patients (50 per group) to account for potential dropouts.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II-III.
* Scheduled for elective, primary, unilateral total knee arthroplasty for osteoarthritis.
* Able to provide written informed consent.

Exclusion Criteria:

* Patient refusal to participate or contraindication to regional anesthesia.
* Known allergy to any study medications (local anesthetics, NSAIDs, tramadol, morphine, paracetamol).
* History of chronic opioid use (defined as daily use for >3 months)
* Pre-existing peripheral neuropathy in the operative limb.
* Severe renal or hepatic insufficiency.
* Cognitive impairment preventing the use of pain scales or questionnaires.
* Revision or bilateral knee arthroplasty.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score with Movement at 24 Hours | 24 and 48. hours postoperatively
  Pain assessed via Numeric Rating Scale (NRS) during active movement (e.g., active knee flexion or straight leg raise). Scale: 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative Pain Scores (Time-Course) | Assessed at 6, 12, and 24 hours postoperatively
  Numeric Rating Scale (NRS) for pain (0-10) assessed at rest and with movement.
Time to First Rescue Analgesia | First 48 postoperative hours
  Time (in minutes) from the end of surgery to the first patient request for rescue tramadol.
Time Up to Go Test | Assessed at 24 hours
  The time taken (in seconds) for the participant to stand up from a standard armchair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. Lower values indicate better functional mobility.
Straight Leg Raise | Postoperative 24. hour
  Assessment of active quadriceps motor function. Defined as the participant's ability to actively lift the operated leg off the bed with the knee fully extended (straight). This will be assessed as a binary outcome (Success = Able to lift unassisted / Failure = Unable to lift).
Knee Range of Motion (ROM) | Baseline (Preoperative) and 24 hours postoperatively
  Active knee flexion (in degrees)
Incidence of Adverse Events | First 48 hours.
  Incidence of postoperative nausea and vomiting (PONV).

CONTACTS AND LOCATIONS:
Overall Officials: Aslan, Principal Investigator — Turgutlu State Hospital

IPD SHARING:
Plan to Share IPD: Yes
All the patient statistics
Supporting Information: SAP, CSR